CLINICAL TRIAL: NCT00244608
Title: A Comparison of the Inflammatory Control of Asthma Provided by One Inhalation of Symbicort® Turbuhaler® 160/4.5 µg/Inhalation b.i.d. Plus As-needed Versus One Inhalation of Symbicort® Turbuhaler® 320/9 µg/Inhalation b.i.d. + One Inhalation of Pulmicort® Turbuhaler® 400 µg/Dose b.i.d. Plus Terbutaline Turbuhaler® 0.4 mg/Inhalation As-needed. A 12-month, Randomised, Double-blind, Parallel-group, Active Controlled, Multinational, Phase IIIB Study in Adult Patients With Asthma, EOS
Brief Title: A Comparison of the Control of Asthma Provided by Symbicort® Turbuhaler® Versus Symbicort® Turbuhaler® Plus Pulmicort® Turbuhaler® Plus Terbutaline Turbuhaler®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5890C00003; EudraCT no. 2004-004042-41
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/Formoterol Turbuhaler
  Other Names: Symbicort
Drug: Budesonide Turbuhaler (Pulmicort)
Drug: Terbutaline Turbuhaler

SUMMARY:
The purpose of this study is to determine if a flexible dose of Symbicort has a similar effect on the airways of patients with asthma as a higher fixed-dose of Symbicort with additional glucocorticosteroids added.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma for at least 6 months
* Prescribed daily use of glucocorticosteroids for at least 3 months prior to visit one

Exclusion Criteria:

* Respiratory infection affecting asthma within 30 days prior to study
* Intake of oral, rectal, or parenteral glucocorticosteroids within 30 days prior to study
* Any significant disease or disorder that may jeopardize the safety of the patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Change in eosinophils in bronchial biopsies (first and last visit) and in sputum (5 times during the 12-month treatment period)

SECONDARY OUTCOMES:
Immunopathology and remodeling in biopsies
Immunopathology and mediators in induced sputum
Severe asthma exacerbations (number of and time to first)
Forced expiratory volume in 1 second (FEV1)
As-needed use
Safety variables, including adverse events and vital signs
All variables assessed over the 12-month treatment period

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (22):
- Denmark (3):
  - Research Site, Aalborg
  - Research Site, Århus C
  - Research Site, Copenhagen
- France (2):
  - Research Site, Montpellier
  - Research Site, Pessac
- Germany (3):
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, Marburg
- Spain (3):
  - Research Site, Baraclado
  - Research Site, Barcelona No. 40
  - Research Site, Barcelona, No. 42
- Sweden (5):
  - Research Site, Gothenburg
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Umeå
  - Research Site, Uppsala
- United Kingdom (6):
  - Research Site, Glasgow
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Southampton